CLINICAL TRIAL: NCT00391066
Title: A Randomized, Open Label, Multicenter, Phase 2 Study to Evaluate the Safety and Efficacy of Lumiliximab in Combination With Fludarabine, Cyclophosphamide, and Rituximab Versus Fludarabine, Cyclophosphamide, and Rituximab Alone in Subjects With Relapsed Chronic Lymphocytic Leukemia
Brief Title: Lumiliximab With Fludarabine, Cyclophosphamide, and Rituximab (FCR) Versus FCR Alone in Subjects With Relapsed Chronic Lymphocytic Leukemia (CLL)
Acronym: LUCID
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 152CL201
Record Dates: First submitted 2006-10-19; First posted 2006-10-23 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2011-04

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: CD23+/CD20+ B-cell CLL; CLL
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Receptors, Fc; lumiliximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): FCR
  F (Fludarabine): 25 mg/m2 daily, every four weeks for 21 weeks
  C (Cyclophosphamide): 250 mg/m2 daily, every four weeks for 21 weeks
  R: (Rituximab): Day 1 50 mg/m2, Day 3 325 mg/m2, for the first week, then single doses of 500 mg/m2 every four weeks, for 21 weeks
  Interventions: Drug: FCR
- 2 (Experimental): FCR + Lumiliximab (L)
  L (Lumiliximab): Day 2 50 mg/m2, Day 4 450 mg/m2, for the first week, then single doses of 500 mg/m2 every four weeks, for 21 weeks.
  F (Fludarabine): 25 mg/m2 daily, every four weeks for 21 weeks
  C (Cyclophosphamide): 250 mg/m2 daily, every four weeks for 21 weeks
  R: (Rituximab): Day 1 50 mg/m2, Day 3 325 mg/m2, for the first week, then single doses of 500 mg/m2 every four weeks, for 21 weeks
  Interventions: Drug: FCR + Lumiliximab

INTERVENTIONS:
Drug: FCR + Lumiliximab — Dose, schedule, and duration specified in the protocol
  Arms: 2
Drug: FCR — Dose, schedule, and duration specified in protocol
  Arms: 1

SUMMARY:
This is a randomized (1:1), open-label, multicenter, active-controlled study in patients with previously treated CD23+ and CD20+ relapsed CLL. Patients will receive treatment with either lumiliximab in combination with FCR or FCR alone.

ELIGIBILITY:
Inclusion Criteria:

* Signed, written EC-approved informed consent form.
* Diagnosis of relapsed CD23+ and CD20+ B cell CLL as defined by NCI WG guidelines.
* Subjects who have received at least 1 but no more than 2 prior single agent or combination treatments for CLL.
* Rai Stage III or IV (Binet Stage C), or Rai Stage I or II (Binet Stage A or B) if determined to have disease progression as evidenced by rapid doubling of peripheral lymphocyte count, progressive lymphadenopathy, progressive splenomegaly, or B symptoms (Staging Criteria - Modified Rai).
* WHO Performance Status less than or equal to 2.
* Age greater than or equal to 18 years.
* Male and female subjects of reproductive potential must agree to follow accepted birth control methods during treatment and for 12 months after completion of treatment.
* Acceptable liver function: bilirubin less than or equal to 2.0 mg/dL (26 µmol/L); AST and ALT less than or equal to 2 times upper limit of normal.
* Acceptable hematologic status: platelet count greater than or equal to 50 x 10^9/L should be unsupported by transfusion; ANC greater than or equal to 1 x 10^9/L.
* Acceptable renal function: creatinine clearance calculated according to the formula of Cockcroft and Gault >50 mL/min; serum creatinine less than or equal to 1.5 times upper limit of normal.

Exclusion Criteria:

* Subjects who are refractory to the following combination therapies: purine analogue + R, purine analogue + C, or purine analogue + CR. Refractory is defined as not achieving at least a PR for a minimum duration of 6 months as determined by treating physician. Purine analogues include fludarabine, pentostatin and cladribine.
* Radiotherapy, radioimmunotherapy, biological therapy, chemotherapy, or other investigational therapy within 4 weeks prior to Study Day 1.
* Previous exposure to lumiliximab or other anti-CD23 antibodies.
* Prior autologous or allogeneic BMT or hematopoetic stem cell transplant.
* Known infection with HIV, hepatitis B, or hepatitis C. Although testing for hepatitis B or hepatitis C is not mandatory, this should be considered for all subjects considered at high risk of hepatitis B or hepatitis C infection and in endemic areas. Subjects with any serological evidence of current or past hepatitis B or hepatitis C exposure are excluded unless the serological findings are clearly due to vaccination.
* Uncontrolled diabetes mellitus.
* Uncontrolled hypertension.
* Transformation to aggressive B-cell malignancy (e.g., large B cell lymphoma, Richter's Syndrome, or PLL).
* Secondary malignancy requiring active treatment (except hormonal therapy).
* Any medical condition that would require long-term use (>1 month) of systemic corticosteroids during study treatment. However, steroid use less than or equal to 1 month is permissible during the study.
* Any serious nonmalignant disease or laboratory abnormality, which in the opinion of the Investigator and/or Sponsor would compromise protocol objectives.
* Active uncontrolled bacterial, viral, or fungal infections.
* New York Heart Association Class III or IV cardiac disease, myocardial infarction within the past 6 months prior to Study Day 1, unstable arrhythmia, or evidence of ischemia on ECG within 30 days prior to Study Day 1.
* Seizure disorders requiring anticonvulsant therapy.
* Severe chronic obstructive pulmonary disease with hypoxemia.
* Major surgery, other than diagnostic surgery, within 4 weeks prior to Study Day 1.
* Clinically active autoimmune disease.
* History of fludarabine-induced autoimmune cytopenia (as judged by the Investigator) or Coombs-positive haemolytic anemia.
* Pregnant or currently breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 627 (Actual)
Dates: Start 2006-11; Primary Completion 2010-07 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Complete Response (CR) rate | Every 3 months until all patients have reached at least week 33

SECONDARY OUTCOMES:
Time to event variables (progression free survival, duration of response, time to next therapy, time to progression and overall survival) | Every 3 months until all patients have reached at least week 33
Response variables | Every 3 months until all patients have reached at least week 33

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (192):
- United States (53):
  - Research Site, Scottsdale, Arizona
  - Research Site, Alhambra, California
  - Research Site, Burbank, California
  - Research Site, Fullerton, California
  - Research Site, La Jolla, California
  - Research Site, Long Beach, California
  - Research Site, Los Angeles, California
  - Research Site, Northridge, California
  - Research Site, Oxnard, California
  - Research Site, Pomona, California
  - Research Site, Redondo Beach, California
  - Research Site, Sacramento, California
  - Research Site, Santa Maria, California
  - Research Site, Fort Myers, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Marietta, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Maywood, Illinois
  - Research Site, Indianapolis, Indiana
  - Research Site, Overland Park, Kansas
  - Research Site, Shreveport, Louisiana
  - Research Site, Boston, Massachusetts
  - Research Site, Detroit, Michigan
  - Research Site, Saint Joseph, Michigan
  - Research Site, Ypsilant,, Michigan
  - Research Site, Minneapolis, Minnesota
  - Research Site, Columbia, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Billings, Montana
  - Research Site, Omaha, Nebraska
  - Research Site, Hackensack, New Jersey
  - Research Site, Morristown, New Jersey
  - Research Site, Chapel Hill, North Carolina
  - Research Site, Raleigh, North Carolina
  - Research Site, Columbus, Ohio
  - Research Site, Kettering, Ohio
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Greenville, South Carolina
  - Research Site, Nashville, Tennessee
  - Research Site, Austin, Texas
  - Research Site, Bedford, Texas
  - Research Site, Dallas, Texas
  - Research Site, Fort Worth, Texas
  - Research Site, Fredericksburg, Texas
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Norfolk, Virginia
  - Research Site, Roanoke, Virginia
  - Research Site, Kennewick, Washington
  - Research Site, Saint Louis, Washington
  - Research Site, Spokane, Washington
  - Research Site, Yakima, Washington
- Argentina (2):
  - Research Site, Córdoba
  - Research Site, Mendoza
- Australia (20):
  - Research Site, Darlinghurst, New South Wales
  - Research Site, Gosford, New South Wales
  - Research Site, St Leonards, New South Wales
  - Research Site, Waratah, New South Wales
  - Research Site, Westmead, New South Wales
  - Research Site, Greenslopes, Queensland
  - Research Site, Herston, Queensland
  - Research Site, South Brisbane, Queensland
  - Research Site, Woolloongabba, Queensland
  - Research Site, Adelaide, South Australia
  - Research Site, Ashford, South Australia
  - Research Site, Woodville, South Australia
  - Research Site, Box Hill, Victoria
  - Research Site, Clayton, Victoria
  - Research Site, East Melbourne, Victoria
  - Research Site, Fitzroy, Victoria
  - Research Site, Freemantle, Western Australia
  - Research Site, Nedlands, Western Australia
  - Research Site, Perth, Western Australia
  - Research Site, Melbourne
- Austria (4):
  - Research Site, Graz
  - Research Site, Innsbruck
  - Research Site, Salzburg
  - Research Site, Vienna
- Belgium (7):
  - Research Site, Antwerp
  - Research Site, Bruges
  - Research Site, Brussels
  - Research Site, Edegem
  - Research Site, Ghent
  - Research Site, Herestraat
  - Research Site, Yvoir
- Brazil (5):
  - Research Site, Goiania - GO
  - Research Site, Porto Alegre
  - Research Site, Rio de Janeiro
  - Research Site, Santo André
  - Research Site, São Paulo
- Canada (8):
  - Research Site, Calgary, Alberta
  - Research Site, Edmonton, Alberta
  - Research Site, Halifax, Nova Scotia
  - Research Site, London, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Hamilton
  - Research Site, Québec
- Czechia (3):
  - Research Site, Brno
  - Research Site, Hradec Králové
  - Research Site, Prague
- France (11):
  - Research Site, Angers
  - Research Site, Bordeaux
  - Research Site, Le Mans
  - Research Site, Lille
  - Research Site, Limoges
  - Research Site, Nantes
  - Research Site, Nice
  - Research Site, Pessac
  - Research Site, Rennes
  - Research Site, Rouen
  - Research Site, Tours
- Germany (6):
  - Research Site, Augsburg
  - Research Site, Dessau
  - Research Site, Frankfurt
  - Research Site, Greifswald
  - Research Site, Kiel
  - Research Site, Würzburg
- Greece (2):
  - Research Site, Athens
  - Research Site, Heraklion
- India (8):
  - Research Site, Ahmedabad
  - Research Site, Bangalore
  - Research Site, Delhi
  - Research Site, Mumbai
  - Research Site, Nashik
  - Research Site, New Delhi
  - Research Site, Pune
  - Research Site, Trivandrum
- Israel (6):
  - Research Site, Ashkelon
  - Research Site, Haifa
  - Research Site, Jerusalem
  - Research Site, Petah Tikva
  - Research Site, Ramat Gan
  - Research Site, Rehovo
- Italy (6):
  - Research Site, Milan
  - Research Site, Novara
  - Research Site, Roma
  - Research Site, Rome
  - Research Site, Rozzano
  - Research Site, Verona
- Research Site, Klaipėda, Lithuania
- New Zealand (5):
  - Research Site, Auckland
  - Research Site, Christchurch
  - Research Site, Hamilton
  - Research Site, Palmerston North
  - Research Site, Wellington
- Poland (7):
  - Research Site, Bialystok
  - Research Site, Gdansk
  - Research Site, Katowice
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Szczecin
  - Research Site, Warsaw
- Portugal (6):
  - Research Site, Almada
  - Research Site, Braga
  - Research Site, Coimbra
  - Research Site, Lisbon
  - Research Site, Porto
  - Research Site, Viseu
- Romania (3):
  - Research Site, Brasov
  - Research Site, Bucharest
  - Research Site, Iași
- Russia (8):
  - Research Site, Nizhny Novgorod
  - Research Site, Obninsk
  - Research Site, Ryazan
  - Research Site, Saint Peterburg
  - Research Site, Saint Petersburg
  - Research Site, Samara
  - Research Site, Saratov
  - Research Site, Yekaterinburg
- Slovakia (3):
  - Research Site, Banská Bystrica
  - Research Site, Bratislava
  - Research Site, Martin
- Spain (6):
  - Research Site, Madrid
  - Research Site, Murcia
  - Research Site, Palma de Mallorca
  - Research Site, Salamanca
  - Research Site, Toledo
  - Research Site, Zaragoza
- United Kingdom (12):
  - Research Site, Bath
  - Research Site, Belfast
  - Research Site, Birmingham
  - Research Site, Bournemouth
  - Research Site, Edinburgh
  - Research Site, Glasgow
  - Research Site, Leeds
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Plymouth
  - Research Site, Surrey
  - Research Site, Taunton

REFERENCES:
- [Background] Byrd JC, Kipps TJ, Flinn IW, Castro J, Lin TS, Wierda W, Heerema N, Woodworth J, Hughes S, Tangri S, Harris S, Wynne D, Molina A, Leigh B, O'Brien S. Phase 1/2 study of lumiliximab combined with fludarabine, cyclophosphamide, and rituximab in patients with relapsed or refractory chronic lymphocytic leukemia. Blood. 2010 Jan 21;115(3):489-95. doi: 10.1182/blood-2009-08-237727. Epub 2009 Oct 20. PMID 19843887
- [Background] Pathan NI, Chu P, Hariharan K, Cheney C, Molina A, Byrd J. Mediation of apoptosis by and antitumor activity of lumiliximab in chronic lymphocytic leukemia cells and CD23+ lymphoma cell lines. Blood. 2008 Feb 1;111(3):1594-602. doi: 10.1182/blood-2007-03-082024. Epub 2007 Nov 21. PMID 18032710
- [Background] Byrd JC, O'Brien S, Flinn IW, Kipps TJ, Weiss M, Rai K, Lin TS, Woodworth J, Wynne D, Reid J, Molina A, Leigh B, Harris S. Phase 1 study of lumiliximab with detailed pharmacokinetic and pharmacodynamic measurements in patients with relapsed or refractory chronic lymphocytic leukemia. Clin Cancer Res. 2007 Aug 1;13(15 Pt 1):4448-55. doi: 10.1158/1078-0432.CCR-06-1463. PMID 17671129
- [Derived] Awan FT, Hillmen P, Hellmann A, Robak T, Hughes SG, Trone D, Shannon M, Flinn IW, Byrd JC; LUCID trial investigators. A randomized, open-label, multicentre, phase 2/3 study to evaluate the safety and efficacy of lumiliximab in combination with fludarabine, cyclophosphamide and rituximab versus fludarabine, cyclophosphamide and rituximab alone in subjects with relapsed chronic lymphocytic leukaemia. Br J Haematol. 2014 Nov;167(4):466-77. doi: 10.1111/bjh.13061. Epub 2014 Aug 8. PMID 25130401